CLINICAL TRIAL: NCT03350815
Title: A Randomized, Double-blind, Parallel-group, Multicenter Study of Secukinumab to Compare 300 mg and 150 mg at Week 52 in Patients With Ankylosing Spondylitis Who Are Randomized to Dose Escalation After Not Achieving Inactive Disease During an Initial 16 Weeks of Open-label Treatment With Secukinumab 150 mg (ASLeap)
Brief Title: Study Estimating the Clinical Difference Between 300 mg and 150 mg of Secukinumab Following Dose Escalation to 300 mg in Patients With Ankylosing Spondylitis
Acronym: ASLeap
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457FUS06
Record Dates: First submitted 2017-10-31; First posted 2017-11-22 (Actual); Results first posted 2022-04-08 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis; ASDAS inactive disease; secukinumab; ASDAS
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: This was a randomized, double-blind, parallel-group, multicenter design which included an initial 16 week open-label period (Treatment Period 1) followed by a randomized, double-blind, parallel-group period (Treatment Period 2),
Who Masked: Participant, Investigator
Masking Description: Patients and Investigators will be blinded to the secukinumab dose during Treatment Period 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Responders (Active Comparator): Patients who achieved an Ankylosing Spondylitis Disease Activity Score (ASDAS) inactive disease (total score <1.3) at both Week 12 and Week 16.
  Interventions: Drug: 150 mg open-label secukinumab; Drug: 150 mg double-blinded secukinumab
- Inadequate responders (Active Comparator): Patients who have active disease, defined as an Ankylosing Spondylitis Disease Activity Score (ASDAS) total score of >1.3 at both Week 12 and Week 16, and who achieved a decrease (improvement) from baseline in total ASDAS score at both Week 12 and Week 16.
  Interventions: Drug: 150 mg open-label secukinumab; Drug: 150 mg double-blinded secukinumab; Drug: 300 mg double-blinded secukinumab
- Non-responders (Active Comparator): Patients who exhibit no change or an increase (worsening) from baseline in total Ankylosing Spondylitis Disease Activity Score (ASDAS) score at either Week 12 or Week 16.
  Non-responders were not entered Treatment Period 2. Non-responders were discontinued from the study at Week 16.
  Interventions: Drug: 150 mg open-label secukinumab

INTERVENTIONS:
Drug: 150 mg open-label secukinumab — All patients in Treatment Period 1 received 150 mg s.c. injection open-label secukinumab.
  Other Names: AIN457
Drug: 150 mg double-blinded secukinumab — Treatment Period 2 Patients who achieved responder status entered Treatment Period 2 and continued to receive 150 mg s.c. (1 s.c. injection of secukinumab 150 mg)
  Other Names: AIN457
  Arms: Inadequate responders; Responders
Drug: 300 mg double-blinded secukinumab — Treatment Period 2 300 mg (2 s.c. injections of the 150 mg dose)
  Other Names: AIN457
  Arms: Inadequate responders

SUMMARY:
This was a study estimating the clinical difference between 300 mg and 150 mg of secukinumab following dose escalation to 300 mg in patients with ankylosing spondylitis

DETAILED DESCRIPTION:
The study used a multicenter design which included an initial 16 week open-label period (Treatment Period 1) followed by a randomized, double-blind, parallel-group period (Treatment Period 2),

1. Screening: A Screening Period took place over 2 separate visits, with the first visit used to assess eligibility and to washout prohibited medications (up to 11 weeks). The second Screening Visit, which occurred at a minimum of 2 weeks prior to the Baseline Visit for all patients, was used to further assess eligibility and to initiate patients on the sensor actigraphy device and morning sleep questionnaires which collected data over the 2-week Screening Period to establish Baseline data. Note: Patients who did not require a washout, and who satisfied all inclusion and none of the exclusion criteria at the first Screening Visit, could initiate the second Screening Visit 1 (SV1) week after their first Screening Visit.
2. Treatment Period 1: Patients who met all of the inclusion criteria and none of the exclusion criteria had a Baseline Visit performed to start Treatment Period 1. During this 16-week period, all patients received open-label secukinumab 150 mg (1 x 1.0mL subcutaneously [s.c.]) at Baseline, Weeks 1, 2, 3, 4, 8, and 12.

At Week 16, patients were placed into 1 of the following groups:

1. Responders (Rs): Patients who achieved ASDAS inactive disease (total score < 1.3) at both Week 12 and Week 16 and who achieved a decrease (improvement) from Baseline in total ASDAS score at both Week 12 and Week 16.
2. Inadequate responders (IRs): Patients who had active disease, defined as an ASDAS total score of ≥ 1.3 at either Week 12 or Week 16, and who achieved a decrease (improvement) from Baseline in total ASDAS score at both Week 12 and Week 16.
3. Nonresponders: Patients who exhibited no change or an increase (worsening) from Baseline in total ASDAS score at either Week 12 or Week 16.

Note: To minimize patient burden, at the Week 16 Visit, the hs-CRP measurement that is part of the ASDAS calculation was imputed from the Week 12 hs-CRP results to allow for assignment into the groups above. Historically, hs-CRP levels have varied little between Week 12 and Week 16 or in previous studies of secukinumab in active AS.

1. Treatment Period 2: Upon completion of the Week 16 visit,

1. Responders entered Treatment Period 2 and continued to receive secukinumab 150 mg every 4 weeks through Week 48 as well as 1 matched placebo dose (s.c. injection) to maintain the integrity of the blind for the randomized IR group.
2. Inadequate responders entered Treatment Period 2 and were randomized (1:1, double blinded) to secukinumab 300 mg or secukinumab 150 mg every 4 weeks through Week 48. Patients knew that they were on secukinumab, but were blinded to dose, so they did not know whether they were receiving 150 mg or 300 mg.
3. Nonresponders were discontinued from the study at Week 16. The only condition that was placed on enrollment targets was that no less than 60% of patients (162 patients) were tumor necrosis factor alpha (TNFα) inhibitor naive (or, no more than 40% of patients were TNF-IR). In theory the percentage of TNFα inhibitor naive patients could have reached 100%, although that was not anticipated.

Patients could discontinue the study at any time. If rescue treatment with prohibited medications (as described in Section 9.4.7) occurred, patients were discontinued from the study and were to return for an End of Study Visit. The End of Study Visit was scheduled approximately 4 weeks after the last study treatment and was performed before any new treatment was initiated. After the End of Study Visit, any serious adverse events (SAEs) that occurred in the following 30 days were required to be reported.

ELIGIBILITY:
Key Inclusion Criteria:

1. Understand and communicate with the investigator, comply with the requirements of the study and give a written, signed and dated informed consent
2. Male or non-pregnant, non-lactating female patients at least 18 years of age
3. Diagnosis of moderate to severe Ankylosing Spondylitis (AS) with prior documented radiologic evidence fulfilling the Modified New York criteria for AS
4. Active AS assessed by total Bath Ankylosing Spondylitis Disease Activity index (BASDAI) ≥ 4 (0-10) at baseline
5. Spinal pain as measured by BASDAI question #2 ≥ 4 cm (0-10 cm) at baseline
6. Total back pain as measured by visual analog scale (VAS) ≥ 40 mm (0-100 mm) at baseline
7. Patients should have been on non-steroidal anti-inflammatory drugs (NSAIDs) at the maximum tolerated dose for at least 4 weeks prior to their Baseline Visit, with an inadequate response or for less than 4 weeks if withdrawn for intolerance, toxicity or contraindications
8. Stable dose of NSAIDs including Cyclooxygenase-1 (COX-1) or Cyclooxygenase-2 (COX-2) inhibitors for at least 2 weeks before their Baseline Visit
9. Patients who have been on a tumor necrosis factor alpha (TNFα) inhibitor (not more than one) must have experienced an inadequate response to previous or current treatment given at an approved dose for at least 3 months prior to baseline or had been intolerant upon administration of an anti-TNFα agent

Key Exclusion Criteria:

1. Total ankylosis of the spine
2. Use of other investigational drugs within 5 half-lives of enrollment, or within 4 weeks before the Baseline Visit, whichever is longer.
3. History of hypersensitivity to any of the study drugs or its excipients or to drugs of similar chemical classes.
4. Chest x-ray, computerized tomography (CT) scan, or chest magnetic resonance imaging (MRI) with evidence of ongoing infectious or malignant process, obtained within 3 months prior to screening and evaluated by a qualified physician.
5. Previous exposure to secukinumab or any other biologic drug directly targeting Interleukin-17 (IL-17), Interleukin-12/23 (IL-12/23), or the IL-17 receptor, or any other biologic immunomodulating agent, except those targeting TNFα
6. Patients who have taken more than one anti-TNFα agent
7. Any intramuscular or intravenous corticosteroid injection within 2 weeks before baseline
8. Any therapy by intra-articular injections (e.g. corticosteroid) within 4 weeks before baseline
9. Previous treatment with any cell-depleting therapies
10. Patients taking high potency opioid analgesics (e.g., methadone, hydromorphone, morphine)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-05-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (63):
- United States (63):
  - Novartis Investigative Site, Jonesboro, Arkansas
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Loma Linda, California
  - Novartis Investigative Site, Palm Desert, California
  - Novartis Investigative Site, Tustin, California
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Aventura, Florida
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Brandon, Florida
  - Novartis Investigative Site, DeLand, Florida
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Plantation, Florida
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Zephyrhills, Florida
  - Novartis Investigative Site, Duluth, Georgia
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Vernon Hills, Illinois
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Monroe, Louisiana
  - Novartis Investigative Site, Cumberland, Maryland
  - Novartis Investigative Site, Hagerstown, Maryland
  - Novartis Investigative Site, Wheaton, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Worcester, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Saint Clair Shores, Michigan
  - Novartis Investigative Site, Edina, Minnesota
  - Novartis Investigative Site, Springfield, Missouri
  - Novartis Investigative Site, Midland Park, New Jersey
  - Novartis Investigative Site, Voorhees Township, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Santa Fe, New Mexico
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Orchard Park, New York
  - Novartis Investigative Site, Potsdam, New York
  - Novartis Investigative Site, Minot, North Dakota
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Dayton, Ohio
  - Novartis Investigative Site, Middleburg Heights, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Corvallis, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Wexford, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Beaumont, Texas
  - Novartis Investigative Site, Colleyville, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Mesquite, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Spokane, Washington
  - Novartis Investigative Site, Charleston, West Virginia
  - Novartis Investigative Site, Manitowoc, Wisconsin
  - Novartis Investigative Site, Onalaska, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Deodhar A, Kivitz AJ, Magrey M, Walsh JA, Mease PJ, Greenwald M, Kianifard F, Elam C, Bommidi GM, Winseck A, Gensler LS. A secukinumab dose-escalation study in patients with ankylosing spondylitis not achieving inactive disease after 16 weeks of treatment. Rheumatology (Oxford). 2025 Apr 1;64(4):1864-1872. doi: 10.1093/rheumatology/keae432. PMID 39133200
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 322 participants were enrolled at 65 sites in the United States
Pre-assignment Details: Of 435 patients screened in the study, 322 (74.0%) completed the Screening phase.
Groups:
- Period 1: Secukinumab 150 mg: Participants received Secukinumab 150 mg in Period 1
- Period 2: Secukinumab 300 mg (Period 1 Inadequate Responders): Participants received Secukinumab 150 mg in Period 1 were assessed as inadequate responders and randomized to receive Secukinumab 300 mg in Period 2
- Secukinumab 150 mg (Period 1 Inadequate Responders): Participants received Secukinumab 150 mg in Period 1 were assessed as inadequate responders and continued with Secukinumab 150 mg in Period 2
- Secukinumab 150 mg (Period 1 Responders): Participants received Secukinumab 150 mg in Period 1 were assessed as responders and continued with Secukinumab 150 mg in Period 2
Period: Period 1
Arm/Group | Period 1: Secukinumab 150 mg | Period 2: Secukinumab 300 mg (Period 1 Inadequate Responders) | Secukinumab 150 mg (Period 1 Inadequate Responders) | Secukinumab 150 mg (Period 1 Responders)
Started | 322 | 0 | 0 | 0
Non-responders (One patient completed Treatment Period 1 and was randomized (secukinumab 150 mg - 300 mg [IR]); however, the patient did not receive any treatment in Treatment Period 2 due to "Technical problems.") | 50 | 0 | 0 | 0
Inadequate Responders | 207 | 0 | 0 | 0
Responders | 22 | 0 | 0 | 0
Completed | 279 | 0 | 0 | 0
Not Completed | 43 | 0 | 0 | 0
Not completed — Adverse Event | 10 | 0 | 0 | 0
Not completed — Technical problems | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 0 | 0 | 0
Not completed — Lack of Efficacy | 15 | 0 | 0 | 0
Not completed — Non-compliance with study treatment | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0 | 0
Period: Period 2
Arm/Group | Period 1: Secukinumab 150 mg | Period 2: Secukinumab 300 mg (Period 1 Inadequate Responders) | Secukinumab 150 mg (Period 1 Inadequate Responders) | Secukinumab 150 mg (Period 1 Responders)
Started | 0 | 102 | 105 | 22
Completed | 0 | 86 | 88 | 22
Not Completed | 0 | 16 | 17 | 0
Not completed — Adverse Event | 0 | 3 | 5 | 0
Not completed — Technical problem | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 4 | 0
Not completed — Lack of Efficacy | 0 | 6 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — New therapy for study indication | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: This is for participants in period 1. 300 mg Arm was not part of Enrollment Set.
Groups:
- Secukinumab 150 mg - 150 mg: AIN457 150 mg - 150 mg
Arm/Group | Secukinumab 150 mg - 150 mg
Number analyzed (Participants) | 322
Age, Categorical [Count of Participants; unit: Participants] — Enrolled Set
  Participants
    <=18 years | 0
    Between 18 and 65 years | 283
    >=65 years | 39
Age, Continuous [Mean (Standard Deviation); unit: Mean] — Enrolled Set
  Mean | 48.02 (13.692)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155
  Male | 167
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Enrolled Set
  Participants
    Caucasian | 284
    Black | 18
    Asian | 11
    Native American | 1
    Pacific Islander | 0
    Other | 3
    Unknown | 5

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants Who Achieved Inactive Disease Based on the Ankylosing Spondylitis Disease Activity Score (ASDAS) Measure
Description: Proportion of participants with inadequate response at week 16 who achieved inactive disease at Week 52 The Ankylosing Spondylitis Disease Activity Score (ASDAS) is a composite index to assess disease activity in AS. The ASDAS-CRP (Ankylosing Spondylitis Disease Activity Score) were utilized to assess the disease activity status.
  * < 1.3 between inactive disease and moderate disease activity,
  * < 2.1 between moderate disease activity and high disease activity, and
  * 3.5 between high disease activity and very high disease activity.
Time Frame: Week 52
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment had been assigned by randomization. According to intent-to-treat principle, patients were analyzed according to the treatment they were assigned to during the randomization procedure.
Measure: Count of Participants; unit: Participants
Groups:
- Secukinumab 150 mg - 300 mg (IR): AIN457 150 mg - 300 mg
- Secukinumab 150 mg - 150 mg (IR): AIN457 150 mg - 150 mg (IR)
Arm/Group | Secukinumab 150 mg - 300 mg (IR) | Secukinumab 150 mg - 150 mg (IR)
Number analyzed (Participants) | 102 | 105
Participants | 9 | 7
Statistical Analysis 1: Comparison: Secukinumab 150 mg - 300 mg (IR) vs Secukinumab 150 mg - 150 mg (IR); Statistical analysis (logistic regression) of ASDAS inactive disease response by visit - in Treatment Period 2 (nonresponder imputation); Test type: Other — Statistical hypothesis tests were not performed for this study; Regression, Logistic — No P value as no hypothesis was tested; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.28 to 2.25]

2. Secondary Outcome: The Proportion of Participants Who Achieved a Clinically Important Improvement on the Ankylosing Spondylitis Disease Activity Score (ASDAS) Scale
Description: A reduction from baseline in ASDAS score of ≥1.1 was considered a clinically important improvement in disease activity in Ankylosing Spondylitis. In this study, ASDAS is used to estimate the difference in response between 150mg and 300mg of secukinumab.
  The Ankylosing Spondylitis Disease Activity Score (ASDAS) is a composite index to assess disease activity in AS. The ASDAS-CRP (Ankylosing Spondylitis Disease Activity Score) wias utilized to assess the disease activity status.
  * < 1.3 between inactive disease and moderate disease activity,
  * < 2.1 between moderate disease activity and high disease activity, and
  * 3.5 between high disease activity and very high disease activity.
Time Frame: Baseline, Week 52
Population: FAS (defined as a patient with inadequte respinse at week 16) for patients with valid assessment for this endpoint.
Measure: Count of Participants; unit: Participants
Groups:
- Secukinumab 150 mg - 300 mg (IR): AIN457 150 mg - 300 mg
  This Arm represents inadequate responders who received 150 mg of the intervention in Period 1 and 2
- Secukinumab 150 mg - 150 mg (IR): AIN457 150 mg - 150 mg
Arm/Group | Secukinumab 150 mg - 300 mg (IR) | Secukinumab 150 mg - 150 mg (IR)
Number analyzed (Participants) | 102 | 105
Participants | 6 | 3
Statistical Analysis 1: Comparison: Secukinumab 150 mg - 300 mg (IR) vs Secukinumab 150 mg - 150 mg (IR); Statistical analysis (logistic regression) of reduction in ASDAS >= 1.1 response by visit - in Treatment Period 2 (nonresponder imputation); Test type: Other — Statistical hypothesis tests were not performed for this study; Regression, Logistic — No P value as no hypothesis was tested; Odds Ratio (OR) = 2.08, 95% CI 2-sided [0.50 to 8.66]

3. Secondary Outcome: Change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: BASDAI is a validated assessment tool using 0 through 10 scales (0 indicating "no problem" and 10 indicating "worst problem"), to characterize six clinical domains pertaining to five major symptoms of AS perceived by the patients. Computed composite scores of 4 or greater indicate suboptimal disease control. In this study, BASDAI is used to estimate the difference in response between 150mg and 300mg of secukinumab.
Time Frame: Baseline, Week 52
Population: FAS for patients with valid assessment for this endpoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Secukinumab 150 mg - 300 mg (IR) | Secukinumab 150 mg - 150 mg
Number analyzed (Participants) | 83 | 85
Score on a scale | 0.18 (0.191) | -0.05 (0.188)
Statistical Analysis 1: Comparison: Secukinumab 150 mg - 300 mg (IR) vs Secukinumab 150 mg - 150 mg; Statistical analysis of total BASDAI change from Week 16 using MMRM - in Treatment Period 2 (FAS); Test type: Other — Statistical hypothesis tests were not performed for this study; Mixed Models Analysis — Least squares means (LSMs) of the treatment groups, LSM treatment difference and 95% confidence interval for treatment difference are from mixed-effects model repeated measures (MMRM) with treatment, visit and TNF-alpha inhibitor status as factors; Least Square Mean of Treatment Differenc = 0.23, 95% CI 2-sided [-0.29 to 0.75], Standard Error of Mean 0.263

4. Secondary Outcome: Proportion of Patients Who Achieved Bath Ankylosing Spondylitis Disease Activity Index 50 (BASDAI-50)
Description: BASDAI-50 represents a change from baseline (improvement) of at least 50% in BASDAI score. In this study, BASDAI is used to estimate the difference in response between 150mg and 300mg of secukinumab.
Time Frame: Baseline, Week 52
Population: FAS for patients with valid assessment for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg - 300 mg (IR) | Secukinumab 150 mg - 150 mg
Number analyzed (Participants) | 102 | 105
Participants | 11 | 9
Statistical Analysis 1: Comparison: Secukinumab 150 mg - 300 mg (IR) vs Secukinumab 150 mg - 150 mg; Statistical analysis (logistic regression) of BASDAI50 response by visit - in Treatment Period 2 (nonresponder imputation) (FAS); Test type: Other — Statistical hypothesis tests were not performed for this study; Regression, Logistic — Odds ratio and 95% confidence interval for odds ratio are from a logistic regression model with treatment (2 treatment groups), TNF-alpha inhibitor status (naive, inadequate responder) and Week 16 body weight (kg) as explanatory variables; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.50 to 3.24]

5. Secondary Outcome: The Proportion of Participants Who Achieved an ASAS 20 Response (Assessment of SpondyloArthritis International Society Criteria)
Description: ASAS 20 response is a validated composite assessment, reflecting the proportion of treated patients who achieve within a defined time frame at least 20% improvement in score in at least 3 of a conventional set of 4 clinical domains relevant to AS and no worsening in the fourth domain. In this study, ASAS20 is used to estimate the difference in response between 150mg and 300mg of secukinumab.
  An ASAS20 response is defined as an improvement of ≥20% from baseline and absolute improvement from baseline of at least 1 on a 0-to-10 scale in at least 3 of the following 4 domains: patient global, total back pain, function (BASFI), and inflammation (average of the last 2 questions of the BASDAI concerning morning stiffness). An absence of deterioration from baseline (deterioration defines as ≥20% worsening and absolute worsening of at last 1 on a 0-to-10 scale) in the potential remaining domain.
Time Frame: Week 52
Population: FAS for patients with valid assessment for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg - 300 mg (IR) | Secukinumab 150 mg - 150 mg
Number analyzed (Participants) | 102 | 105
Participants | 19 | 22
Statistical Analysis 1: Comparison: Secukinumab 150 mg - 300 mg (IR) vs Secukinumab 150 mg - 150 mg; Statistical analysis (logistic regression) of BASDAI20 response by visit - in Treatment Period 2 (nonresponder imputation) (FAS); Test type: Other — Statistical hypothesis tests were not performed for this study; Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.43 to 1.73]

6. Secondary Outcome: The Proportion of Participants Who Achieved an ASAS 40 Response
Description: ASAS 40 response is a validated composite assessment, reflecting the proportion of treated patients who achieve within a defined time frame at least 40% improvement in score in at least 3 of a conventional set of 4 clinical domains relevant to AS and no worsening in the fourth domain. In this study, ASAS40 is used to estimate the difference in response between 150mg and 300mg of secukinumab.
  An ASAS40 response is defined as a ≥40% improvement in 3 of the 4 domains with an absolute improvement of at least 2 on a 0-to-10 scale, and no worsening in the remaining domain.
Time Frame: Week 52
Population: FAS for patients with valid assessment for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg - 300 mg (IR) | Secukinumab 150 mg - 150 mg
Number analyzed (Participants) | 102 | 105
Participants | 10 | 8
Statistical Analysis 1: Comparison: Secukinumab 150 mg - 300 mg (IR) vs Secukinumab 150 mg - 150 mg; Statistical analysis (logistic regression) of ASAS40 response by visit - in Treatment Period 2 (nonresponder imputation) (FAS); Test type: Other — Statistical hypothesis tests were not performed for this study; Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.49 to 3.46]

7. Secondary Outcome: The Proportion of Patients Who Achieved an ASAS Partial Remission
Description: The ASAS partial remission criteria are defined as a value not above 2 units in each of the four main domains on a scale of 0-10. In this study, ASAS partial remission is used to estimate the difference in response between 150mg and 300mg of secukinumab.
Time Frame: Week 52
Population: FAS for patients with valid assessment for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg - 300 mg (IR) | Secukinumab 150 mg - 150 mg
Number analyzed (Participants) | 102 | 105
Participants | 12 | 12
Statistical Analysis 1: Comparison: Secukinumab 150 mg - 300 mg (IR) vs Secukinumab 150 mg - 150 mg; Statistical analysis (logistic regression) of ASAS partial remission response by visit - in Treatment Period 2 (nonresponder imputation) (FAS); Test type: Other — Statistical hypothesis tests were not performed for this study; Regression, Logistic — Odds ratio and 95% confidence interval for odds ratio are from a logistic regression model with treatment (2 treatment groups), TNF-alpha inhibitor status(naive, inadequate responder) and Week 16 body weight (kg) as explanatory variables; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.44 to 2.41]

8. Secondary Outcome: Change in ASAS - Health Index Over Time
Description: The ASAS-HI is a self-administered questionnaire and measures functioning and health over 17 aspects of health and 9 environmental factors in patients with spondyloarthritis. Patients score each item as "I agree" and "I do not agree". In this study, ASAS-HI is used to estimate the difference in response between 150mg and 300mg of secukinumab. Lower score indicating a better health status
Time Frame: Baseline, Week 52
Population: FAS for patients with valid assessment for this endpoint.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Secukinumab 150 mg - 300 mg (IR) | Secukinumab 150 mg - 150 mg
Number analyzed (Participants) | 83 | 85
scores on a scale | 0.51 (0.320) | 0.38 (0.315)
Statistical Analysis 1: Comparison: Secukinumab 150 mg - 300 mg (IR) vs Secukinumab 150 mg - 150 mg; Statistical analysis of change from Week 16 in ASAS-Health Index using MMRM by visit - in Treatment Period 2 (FAS); Test type: Other — Statistical hypothesis tests were not performed for this study; Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.74 to 1.01]

9. Secondary Outcome: Change in Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue Over Time
Description: Fatigue was assessed using the 13-item FACIT-fatigue scale for the assessment of fatigue in cancer patients.24 The FACIT-Fatigue is a validated questionnaire that was originally developed for the precise evaluation of fatigue levels in cancer patients with anemia. It consists of 13 questions using a 5 point scale (0=not at all; 1 = a little bit, 2 = somewhat, 3 = quite a bit and 4 = very much). Responses to each question were added with equal weight to obtain a total score. The range of possible scores is 0-52, with 0 corresponding to the highest level of fatigue and 52 corresponding to the lowest level of fatigue.
Time Frame: Baseline, Week 52
Population: FAS for patients with valid assessment for this endpoint.
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | Secukinumab 150 mg - 300 mg (IR) | Secukinumab 150 mg - 150 mg
Number analyzed (Participants) | 83 | 85
Score | -1.93 (0.954) | -0.92 (0.938)
Statistical Analysis 1: Comparison: Secukinumab 150 mg - 300 mg (IR) vs Secukinumab 150 mg - 150 mg; Test type: Other — Statistical hypothesis tests were not performed for this study; Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-3.62 to 1.61]

ADVERSE EVENTS:
Time Frame: AEs were collected from first dose of study treatment until end of study treatment at week 52
Description: Adverse Events (AEs) are any untoward sign or symptom that occurs during the study treatment and up to 52 weeks
Groups:
- Treatment Period 2 Secukinumab 150 mg - 150 mg (R): Treatment Period 2 Secukinumab 150 mg - 150 mg (R)
- Treatment Period 1 Secukinumab 150 mg: Treatment Period 1 Secukinumab 150 mg
- Treatment Period 2 Secukinumab 150 mg - 300 mg (IR): Treatment Period 2 Secukinumab 150 mg - 300 mg (IR)
- Treatment Period 2 Secukinumab 150 mg - 150 mg (IR): Treatment Period 2 Secukinumab 150 mg - 150 mg (IR)
Arm/Group | Treatment Period 2 Secukinumab 150 mg - 150 mg (R) | Treatment Period 1 Secukinumab 150 mg | Treatment Period 2 Secukinumab 150 mg - 300 mg (IR) | Treatment Period 2 Secukinumab 150 mg - 150 mg (IR)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/322 | 0/101 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/22 | 11/322 | 7/101 | 3/105
Other Adverse Events (participants affected / at risk) | 7/22 | 50/322 | 30/101 | 32/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period 2 Secukinumab 150 mg - 150 mg (R) (N=22) | Treatment Period 1 Secukinumab 150 mg (N=322) | Treatment Period 2 Secukinumab 150 mg - 300 mg (IR) (N=101) | Treatment Period 2 Secukinumab 150 mg - 150 mg (IR) (N=105)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period 2 Secukinumab 150 mg - 150 mg (R) (N=22) | Treatment Period 1 Secukinumab 150 mg (N=322) | Treatment Period 2 Secukinumab 150 mg - 300 mg (IR) (N=101) | Treatment Period 2 Secukinumab 150 mg - 150 mg (IR) (N=105)
Diarrhoea (Gastrointestinal disorders) | 0 | 18 | 7 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 15 | 6 | 8
SARS-CoV-2 test negative (Investigations) | 2 | 2 | 7 | 8
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 15 | 6 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6 | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT03350815/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT03350815/SAP_001.pdf